CLINICAL TRIAL: NCT03496701
Title: Performance of Wearers of MyDay Sphere Lenses After A Refit With MyDay Energys Lenses for One Week
Brief Title: Performance of Wearers of Stenfilcon A Contact Lenses After A Refit With Test Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-86
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Stenfilcon A / Test lens (Experimental): All subjects will first wear stenfilcon A contact lenses for one week, then refitted with test contact lenses to wear for one week.
  Interventions: Device: Test lens; Device: control lens

INTERVENTIONS:
Device: Test lens — contact lens
  Other Names: stenfilcon A Test lens
Device: control lens — contact lens
  Other Names: stenfilcon A Control lens

SUMMARY:
The aim of this study is to determine if habitual or adapted wearers of stenfilcon A control contact lenses can be refit into test lenses and be successful after one week of daily wear.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, open label, bilateral, daily wear, one week dispensing study comparing performance of wearers of stenfilcon A control contact lenses after refit with test contact lenses.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 35 years of age (inclusive)
* Has read and signed the informed consent letter
* Is willing and anticipated to follow instructions and maintain the appointment schedule
* Habitually wears soft spherical contact lenses with a power between -1.00D to -6.00D (inclusive) for a minimum 5 days per week, 10 hours per day and anticipates no difficulty wearing contact lenses for 7 days per week, 10 hours per day.
* Habitually wears or is able to be adequately refit into MyDay Sphere lenses
* Demonstrates an acceptable fit with the study lenses
* Is correctable to a distance visual acuity of 0.20 logMAR (approximately 20/30) or better (in each eye) with the study contact lenses
* Uses digital devices, (e.g. computer, tablet, smart phone, iPad), for more than 4 hours a day, 5 days a week.
* Manifest cylindrical spectacle refraction does not exceed -0.75DC in either eye
* Has clear corneas and no active ocular disease
* Has a contact lens refraction that fits within the available parameters of the study lenses.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Is participating in any concurrent clinical research study
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a systemic condition that, in the opinion of the investigator, may affect the study measures
* Is using any systemic or topical medications that in the opinion of the investigator may affect the study measures.
* Presents with slit lamp findings or clinically significant anterior segment abnormalities that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Significant pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (or history in past year)
  * Seborrheic eczema of eyelid region, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study
* Has aphakia, keratoconus or a highly irregular cornea.
* Has presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone refractive surgery.
* Is pregnant, lactating or planning a pregnancy (by verbal communication) at the time of enrollment
* Has participated in any other type of eye related clinical or research study within the last 7 days
* Is habitually using rewetting/ lubricating eye drops (more than once per day)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ardaya, Principal Investigator — Golden Optometric Group, CA; Shane Kannarr, Principal Investigator — Kannarr Eye Care, KS; Michael Cymbor, Principal Investigator — Nittany Eye Associates, PA; Wayne Golden, Principal Investigator — Golden Vision, FL; Eric M. White, Principal Investigator — CA
Locations (4):
- United States (4):
  - Eric White, O.D., Inc., San Diego, California
  - Golden Optometric Group, Whittier, California
  - Golden Vision, Sarasota, Florida
  - Nittany Eye Associates, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: All subjects will first wear stenfilcon A contact lenses for one week, then refitted with test contact lenses to wear for one week.
  Test lens: contact lens
  control lens: contact lens
Period: Overall Study
Arm/Group | Overall Study
Started | 77
Completed | 77
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Fit Acceptance
Description: Overall lens fit acceptance on a scale of 0-4, 0.5 steps (Scale: 0=should not be worn, 4=perfect)
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stenfilcon A Test Lens: All subjects will first wear stenfilcon A test contact lenses for one week.
  stenfilcon A test lens: contact lens
- Stenfilcon A Control Lens: All subjects will first wear stenfilcon A control contact lenses for one week.
  stenfilcon A control lens: contact lens
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
units on a scale | 3.90 (0.26) | 3.81 (0.34)

2. Primary Outcome: Overall Lens Fit Acceptance
Description: Overall lens fit acceptance on a scale of 0-4, 0.5 steps (Scale: 0=should not be worn, 4=perfect)
Time Frame: 1 week on each study lenses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
units on a scale | 3.79 (0.47) | 3.83 (0.35)

3. Secondary Outcome: Lens Centration
Description: Lens centration was assessed on a 3 point scale (1-Optimum, 2- Decentration acceptable, 3-Decentration unacceptable)
Time Frame: Baseline - After 10 minutes of lens dispense
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
Participants
  Optimum | 76 | 76
  Acceptable | 1 | 1
  Unacceptable | 0 | 0

4. Secondary Outcome: Lens Centration
Description: Lens centration was assessed on a 3 point scale (1-Optimum, 2- Decentration acceptable, 3-Decentration unacceptable)
Time Frame: 1 week on each study lenses
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
Participants
  Optimum | 75 | 76
  Acceptable | 2 | 1
  Unacceptable | 0 | 0

5. Secondary Outcome: Post-blink Movement
Description: Post-blink movement assessed on a scale of 0-4, 1 step size (Scale: 0=Insufficient, 1=Minimal, 2=Optimal, 3=Moderate, 4=Excessive)
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
units on a scale | 2.04 (0.34) | 1.97 (0.36)

6. Secondary Outcome: Post-blink Movement
Description: as for outcome 5
Time Frame: 1 week on each study lenses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 77 | 77
units on a scale | 1.92 (0.42) | 1.96 (0.34)

ADVERSE EVENTS:
Time Frame: From dispense up to 1 week on each study lenses, a total of 2 weeks.
Arm/Group | Stenfilcon A Test Lens | Stenfilcon A Control Lens
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT03496701/Prot_SAP_001.pdf